CLINICAL TRIAL: NCT02328339
Title: Forearm Blood Flow Response to Acute Consumption of Black Tea
Brief Title: Tea and Forearm Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REF-BEV-1797
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Vascular Function
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black tea (Experimental): Approximately 400 mg total polyphenols in 240 ml hot water (loading dose; 2 hours before the start of measurements; t=0) and 130 mg total polyphenols in 120 ml hot water (maintenance dose just before start of the measurements; t=120 min)
  Interventions: Other: Tea
- Placebo (Placebo Comparator): Caramel colour, maltodextrin and tea flavour in 240 ml hot water (2 hours before the start of measurements; t=0) and 120 ml hot water (maintenance dose just before start of the measurements; t=120 min)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tea — Black tea infusion equivalent to approximately 530 mg total polyphenols expressed as gallic acid equivalents
  Arms: Black tea
Other: Placebo — Placebo matched to tea with respect to taste and appearance
  Arms: Placebo

SUMMARY:
The study will explore the benefit of tea for microcirculation. Subjects will consume tea ar a placebo matched for taste and appearance in a blinded cross over design.

DETAILED DESCRIPTION:
Epidemiological studies indicate that regular consumption of black tea reduces the risk of cardiovascular diseases. Tea consumption can result in improvements in endothelial function of conduit arteries as measured by flow mediated dilation.

Less is known however about its effects in other vascular beds. The study will test the hypothesis that tea affects endothelial function in the muscle microcirculation. This will be done by assessment of forearm blood flow using venous occlusion plethysmography after consumption of black tea against or placebo in a randomised, full cross-over study in 20 healthy middle-aged to elderly subjects

ELIGIBILITY:
Inclusion Criteria:

* Males and post menopausal (> 1 years) females
* Aged ≥ 45 and ≤ 75 years
* Body mass index (BMI) of ≥ 18.0 and ≤ 35.0 kg/m2
* Judged to be in good health on the basis of medical history, physical examination and routine laboratory tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, glucose, highly sensitive C-reactive protein).
* Normal blood coagulation as assessed by routine lab tests

Exclusion Criteria:

* Strenuous exercise > 2 hours per week. Strenuous exercise is defined as exercise which induces sweating and causes sufficient breathlessness to limit conversation
* Current smoker or has stopped smoking less than 6 months before start of study
* Self reported alcohol intake of > 21 units/week)
* Established cardiovascular disease or clinically significant arrhythmia
* Diabetes mellitus
* Blood pressure > 160/100 mmHg
* Taking medication that might affect endothelial function (as judged by the PI)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow response to acetylcholine | During acetylcholine infusion 120-140 min after first tea/placebo intake
  Does tea ingestion change mean forearm blood flow response to acetylcholine when compared to placebo

SECONDARY OUTCOMES:
Forearm blood flow response to sodium nitropusside | During sodium nitropusside infusion 170-190 min after first tea/placebo intake
  Does tea ingestion change mean forearm blood flow response to sodium nitropusside when compared to placebo
Forearm blood flow response to L-NMMA | During L-NMMA infusion 220-240 min after first tea/placebo intake
  Does tea ingestion change mean forearm blood flow response to L-NG-monomethyl Arginine (L-NMMA) when compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sean Roerink, Dr., Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Derived] Greyling A, Wolters TLC, de Bresser DM, Roerink SHPP, Riksen NP, Mulder TP, Rowson MJ, Hopman MT, Thijssen DHJ. The acute effect of black tea consumption on resistance artery endothelial function in healthy subjects. A randomized controlled trial. Clin Nutr ESPEN. 2018 Feb;23:41-47. doi: 10.1016/j.clnesp.2017.10.011. Epub 2017 Nov 8. PMID 29460812